CLINICAL TRIAL: NCT02666092
Title: Protists and Nematodes Fish Parasites: From Their Circulation in Ecosystems to Their Impact on Human Health - Role of Anisakidae and/or Fish Flesh Antigens in Fish Allergies.
Brief Title: Anisakis Blastocystis Cryptosporidium Fish Serology
Acronym: ABCFish2
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Institut Pasteur de Lille (Other); ANSES (Other); Hôpital Cochin (Other); Région Nord-Pas de Calais, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_43; 2014-A00855-42 (Other: ID RCB number, ANSM)
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Allergy to Fish; Allergy; Anisakis
Keywords: IgE; Immunoelectrophoresis; Western Blot; ImmunoCAP
MeSH Terms: conditions — Hypersensitivity; Anisakiasis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Fish allergy: 51 subjects presenting allergic manifestations after digestive, cutaneous, or respiratory contact with fish will be recruited.
  Interventions will include:
  * A questionnaire on domestic exposure to fish, and on the characteristics of clinical manifestations
  * A detection of anti-Anisakis and anti-fish antibodies
  Interventions: Other: Questionnaire; Biological: Detection of anti-Anisakis and anti-fish antibodies
- Control: 51 subjects presenting no allergic manifestations after contact with fish.
  Interventions will include:
  * A questionnaire on domestic exposure to fish
  * A detection of anti-Anisakis and anti-fish antibodies
  Interventions: Other: Questionnaire; Biological: Detection of anti-Anisakis and anti-fish antibodies

INTERVENTIONS:
Other: Questionnaire — Questionnaire on domestic exposure to fish, and, for patients with fish allergy, on the characteristics of clinical manifestations)
Biological: Detection of anti-Anisakis and anti-fish antibodies — Anti-fish IgE will be detected using ImmunoCAP. Anti-Anisakis antibodies will be detected using ImmunoCAP (IgE), immunoelectrophoresis (precipitins) and Western Blot.

SUMMARY:
Anisakidae frequently infect fish species that are commonly eaten by humans. Some of them are recognized as zoonotic diseases agents, and have a high impact on human health.

Infestation results from the ingestion of living larvae from contaminated fishes. It can be asymptomatic or symptomatic, resulting in acute gastric, acute intestinal or chronic forms. Allergic manifestations are frequently encountered in gastric forms, but allergic symptoms can also occur in isolation, after ingestion of Anisakidae antigens contained in raw or cooked fish, and may masquerade as fish allergy.

In this study, we aim to characterize the relationship between Anisakidae and/or fish sensitization and the presence of allergic manifestations in patients recruited in the general population and presenting fish allergy resulting from ingestion, cutaneous or respiratory contact. We will also determine the respective role of Anisakidae or fish sensitization in patients with fish allergy. Then, we will determine the prevalence of previous Anisakidae infections among these patients and a matched control population. We will also compare the performances of serological tests (ImmunoCAP, immunoelectrophoresis and Western Blot) for the diagnosis of Anisakidae allergy or infection. Lastly, we will explore the relationship between domestic exposure to Anisakidae or fish antigens and the occurrence of associated pathologies (Anisakidae or fish allergy/sensitization; Anisakidae infection).

DETAILED DESCRIPTION:
First, 51 patients with fish allergy will be recruited from the Parasitology-Mycology and Immunology Laboratories of Lille University Hospital databases (serology for anti-Anisakis or anti-fish detection). Then, clinical (characteristics of allergic manifestations) and epidemiological (domestic exposure to fish) data will be collected, and anti-fish or Anti-Anisakis antibodies will be detected using ImmunoCAP (IgE), or ImmunoCAP, immunoelectrophoresis, Western Blot, respectively. Similar serological tests will be performed for a control group of 51 matched subjects who will be recruited among Lille University Hospital workers.

ELIGIBILITY:
Inclusion Criteria:

ALLERGIC PATIENTS:

* Previous serological assessment for anti-Anisakis or anti-fish antibodies detection (ImmunoCap and/or immunoelectrophoresis) in Lille University Hospital Center, and volume of serum conserved ≥500 µl
* Allergic manifestations after contact with fish (asthma, allergic rhinitis, conjunctivitis, chronic or acute urticaria, dermatitis/eczema, eosinophilic gastroenteritis, gingivostomatitis, angioedema, bronchospasm, anaphylaxis)

CONTROL SUBJECTS:

* Serological assessment for infectious disease during a routine occupational health consultation in Lille University Hospital Center
* Absence of fish allergy

Exclusion Criteria:

* Pregnant or breast-feeding female
* Patient with no social insurance
* Patient unwilling to comply with the protocol
* Patient unable to understand the study and its objectives
* Patient under guardianship

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The recruited population will include:
  * 51 patients with fish allergy
  * 51 matched control subjects (sex, age +/- 5 years)
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2015-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
the frequency of anti-Anisakis and/or anti-fish IgE by serum analysis | contact by phone during 30 min at only visit (inclusion)
  comparison between subjects with fish allergy and a matched control population, presenting no fish allergy.

SECONDARY OUTCOMES:
anti-Anisakis and/or anti-fish IgE level by serum analysis | contact by phone during 30 min at only visit (inclusion)
  Comparison between subjects with fish allergy and a matched control population, presenting no fish allergy.
the frequency of anti-Anisakis and anti-fish IgE in patients with fish allergy by serum analysis | contact by phone during 30 min at only visit (inclusion)
nomber of subjects of previous Anisakidae infections | contact by phone during 30 min at only visit (inclusion)
  questionnaire-based diagnosis, supported by serological testing between patients with fish allergy and a matched control population, presenting no fish allergy.
Measure of the performances of serological tests | at work medical visit (inclusion)
  Comparison of the performances of serological tests (ImmunoCAP, immunoelectrophoresis and Western Blot) for the diagnosis of Anisakidae allergy or infection.
The frequency of domestic exposure to fish parasites antigens by questionnaire | contact by phone during 30 min at only visit (inclusion)
  It will be compared between Anisakis or fish allergic/sensitized subjects and non-allergic/non sensitized subjects.
  It will be compared between patients with or without previous Anisakidosis. Fish exposure will be determined taking into account the handled fish species and the local prevalences of fish parasites.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel DUTOIT, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU, Lille, France

IPD SHARING:
Plan to Share IPD: No